CLINICAL TRIAL: NCT00527514
Title: A Prospective, Open-label Study to Assess the Efficacy and Safety of an Olmesartan and Amlodipine Based Treatment Regimen in Subjects With Stage 1 and Stage 2 Hypertension
Brief Title: Blood Pressure Lowering Ability and Safety of an Olmesartan and Amlodipine Based Treatment Regimen in Patients With Stage I and Stage II Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: William Waverczak, Daiichi Sankyo
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8663-402
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Results first posted 2009-09-23 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Hypertension
Keywords: Hypertension; Angiotensin Receptor Blocker; Calcium Channel Blocker; Stage I and II Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Olmesartan Medoxomil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Amlodipine; Drug: Olmesartan medoxomil plus amlodipine

INTERVENTIONS:
Drug: Amlodipine — Tablets
Drug: Olmesartan medoxomil plus amlodipine — Tablets

SUMMARY:
This study will be conducted to assess the efficacy and safety of an amlodipine/olmesartan treatment regimen in stage 1 and stage 2 hypertensive subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males or females greater than or equal to 18 years of age
* Patients with a mean seated systolic blood pressure (MSSBP) greater than or equal to 140 mm Hg but less than or equal to 199 mm Hg or a mean seated diastolic blood pressure (MSDBP) greater than or equal to 90 mm Hg and less than or equal to 109 mm Hg, following a period of taking only placebo
* Patients with a mean daytime (8AM-4PM) systolic blood pressure greater than or equal to 135 mm Hg and less than or equal to 199 mm Hg and a mean daytime diastolic blood pressure less than or equal to 109 mm Hg as measured by an ambulatory blood pressure monitoring device (ABPM), after a period of taking only placebo
* If female, must have negative serum pregnancy test at screening and be either post-menopausal (greater than or equal to 1 year), had a hysterectomy or tubal ligation at least 6 months before consent or if of childbearing potential, must practice approved measures of birth control throughout study

Exclusion Criteria:

* History of stroke or transient ischemic attack (TIA) within the last one year
* History of myocardial infarction, coronary angioplasty, coronary artery bypass graft, or heart failure within the past 6 months
* Patients with secondary hypertension of any etiology, such as renal disease, pheochromocytoma, or Cushing's syndrome
* Type I diabetes. Patients with Type II diabetes on stable treatment, with fasting glucose <160 mg/dl may enroll
* Patients with hemodynamically significant cardiac valvular disease
* Patients with clinically significant cardiac conduction defects, including second or third degree AV block, left bundle branch block, sick sinus syndrome, atrial fibrillation, atrial flutter, an accessory bypass tract, or any arrhythmia requiring medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Buena Park, California
  - Long Beach, California
  - Los Angeles, California
  - Sacramento, California
  - Tustin, California
  - Westlake Village, California
  - Castle Rock, Colorado
  - Pembroke Pines, Florida
  - Orland Park, Illinois
  - Natick, Massachusetts
  - New York, New York
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Beaver, Pennsylvania
  - Greer, South Carolina
  - Carrolton, Texas
  - Corpus Christi, Texas
  - Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 18 US sites over 4 months (September 2007 to December 2007) from each physician's clientele base. Approximately 150 eligible participants, men and women at least 18 years of age with hypertension or uncontrolled hypertension on current medication, were to receive active treatment
Pre-assignment Details: After placebo treatment, participants with a mean systolic blood pressure (SBP)≥140 mmHg and ≤199 mmHg or a mean diastolic BP (DBP)≥90 and ≤109 mmHg with a difference between mean SBPs ≤15 mmHg and a mean 8-hr daytime SBP of ≥135 mmHg and ≤199 mmHg, and mean 8-hr daytime DBP of <110 mmHg by ambulatory BP monitoring were considered eligible.
Groups:
- Amlodipine and Olmesartan, if Necessary: All eligible participants began the active treatment period with amlodipine (Aml) 5 mg for Weeks 1-3. If blood pressure was greater than 120/80 at the end of 3 weeks, participants were titrated to the next regimen for weeks 4-6, and so on for weeks 7-9 and 10-12.
Period: Weeks 1-3: Amlodipine (Aml) 5mg
Arm/Group | Amlodipine and Olmesartan, if Necessary
Started | 185
Completed | 184 (1 participant dropped out. 2 participants were subsequently mis-titrated to the third regimen.)
Not Completed | 1
Not completed — Adverse Event | 1
Period: Weeks 4-6: Aml 5mg+Olmesartan 20 mg
Arm/Group | Amlodipine and Olmesartan, if Necessary
Started | 180 (184 -2 who were mis-titrated -2 who met blood pressure goal = 180)
Completed | 178
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Weeks 7-9: Aml 5 mg + Olmesartan 40 mg
Arm/Group | Amlodipine and Olmesartan, if Necessary
Started | 161 (178 -19 who met blood pressure goal + 2 who were mis-titrated = 161)
Completed | 158
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Period: Weeks 10-12:Aml 10 mg +Olmesartan 40 mg
Arm/Group | Amlodipine and Olmesartan, if Necessary
Started | 134 (158 -24 who met blood pressure goal = 134)
Completed | 132
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Amlodipine and Olmesartan, if Necessary: Week 1-3 all participants: Amlodipine 5mg; Week 4-6 Amlodipine 5 mg/olmesartan 20 mg if mean SBP >= 120/80 mm Hg; Week 7-9 Amlodipine 5 mg/ olmesartan 40 mg if mean SBP >= 120/80 mm Hg; Week 10-12 Amlodipine 10 mg/olmesartan 40 mg if mean SBP >= 120/80 mm Hg
Arm/Group | Amlodipine and Olmesartan, if Necessary
Number analyzed (Participants) | 185
Age Continuous [Mean (Standard Deviation); unit: years] | 56.8 (9.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 105
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 14
  Black or African American | 26
  White | 144
  American Indian or Alaska Native | 1
Region of Enrollment [Number; unit: participants]
  United States | 185
Stage of Hypertension [Number; unit: Participants] — Stage I hypertension is defined as systolic blood pressure (SBP) of 140 - 159 mmHg and diastolic blood pressure (DBP) of 90 - 99 mmHg; Stage II is defined as SBP ≥ 160 mmHg or DBP ≥ 100 mm Hg.
  Participants
    Stage 1 | 82
    Stage 2 | 103
24-Hour Ambulatory Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 85.8 (7.91)
24-hour Ambulatory Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 144.6 (10.88)
Heart Rate [Mean (Standard Deviation); unit: beats/minute] | 75.1 (10.82)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — Seated cuff measurement as opposed to ambulatory measurement.
  mm Hg | 158.2 (12.63)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean 24-hour Systolic Blood Pressure Measured by Ambulatory Monitoring
Time Frame: Baseline to 12 Weeks
Population: The ambulatory blood pressure monitoring (ABPM) subset were subjects who received at least one dose of active study medication and had a baseline ABPM and end of study ABPM measurement.This = 172 participants.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Overall Active Treatment Period
Number analyzed (Participants) | 172
mm Hg | -21.4 (0.80)
Statistical Analysis 1: Comparison: Overall Active Treatment Period; The sample size of this study was not based on the statistical power consideration and was considered as sufficient for the evaluation of the efficacy and safety of the proposed olmesartan medoxomil-based treatment regimen; Test type: Superiority or Other; p < 0.0001, one-sample t-test — No multiplicity adjustments

2. Secondary Outcome: Change From Baseline in Daytime and Nighttime Ambulatory Systolic Blood Pressure
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Overall Active Treatment Period
Number analyzed (Participants) | 172
mm Hg
  Daytime | -23.1 (0.92)
  Nighttime | -18.5 (0.91)
Statistical Analysis 1: Comparison: Overall Active Treatment Period; Statistical analysis parameters apply to both the daytime and nighttime rows; Test type: Superiority or Other; p < 0.0001, One-sample t-test — No multiplicity adjustments

3. Secondary Outcome: Change From Baseline in Cuff Systolic Blood Pressure for the Amlodipine 5mg Group.
Description: Change from study baseline in cuff systolic pressure (as measured by an Omron device) to the end of the treatment period. The Last Observation Carried Forwarded (LOCF) approach was used for the analysis.
Time Frame: Baseline to end of week 3
Population: ITT (efficacy cohort)
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Group 1 Amlodipine 5 mg: All participants started the Active Treatment period with 5 mg of amlodipine for 3 weeks.
Arm/Group | Group 1 Amlodipine 5 mg
Number analyzed (Participants) | 185
mm Hg | -10.1 (0.97)
Statistical Analysis 1: Comparison: Group 1 Amlodipine 5 mg; Test type: Superiority or Other; p < 0.0001, One-sample t-test — No multiplicity adjustments

4. Secondary Outcome: Change From Baseline in Cuff Systolic Blood Pressure for the Amlodipine 5mg + Olmesartan 20 mg Group.
Description: as for outcome 3
Time Frame: Baseline to end of week 6
Population: ITT (efficacy cohort)
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Group 2 - Aml 5 mg + Olmesartan 20 mg: Participants from Group 1 who did not meet the blood pressure goal after 3 weeks were titrated to Aml 5 mg + olmesartan 20 mg.
Arm/Group | Group 2 - Aml 5 mg + Olmesartan 20 mg
Number analyzed (Participants) | 179
mm Hg | -18.0 (0.92)
Statistical Analysis 1: Comparison: Group 2 - Aml 5 mg + Olmesartan 20 mg; Test type: Superiority or Other; p < 0.0001, one-sample t-test — No multiplicity adjustments

5. Secondary Outcome: Change From Baseline in Cuff Systolic Blood Pressure for the Amlodipine 5mg + Olmesartan 40 mg Group
Description: as for outcome 3
Time Frame: Baseline to end of week 9
Population: ITT (efficacy cohort)
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Group 3 - Aml 5 mg + Olm 40 mg: Participants from Group 2 who did not meet the blood pressure goal after 3 weeks were titrated to Aml 5 mg + olmesartan 40mg.
Arm/Group | Group 3 - Aml 5 mg + Olm 40 mg
Number analyzed (Participants) | 160
mm Hg | -20.5 (1.01)
Statistical Analysis 1: Comparison: Group 3 - Aml 5 mg + Olm 40 mg; Test type: Superiority or Other; p < 0.0001, One-sample t-test — No multiplicity adjustments

6. Secondary Outcome: Change From Baseline in Cuff Systolic Blood Pressure for the Amlodipine 10 mg + Olmesartan 40 mg Group
Description: as for outcome 3
Time Frame: Baseline to end end of week 12
Population: ITT (efficacy cohort)
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Group 4 - Aml 10 mg + Olm 40 mg
Number analyzed (Participants) | 133
mm Hg | -24.6 (1.18)
Statistical Analysis 1: Comparison: Group 4 - Aml 10 mg + Olm 40 mg; Test type: Superiority or Other; p < 0.0001, one-sample t-test — No multiplicity adjustments

ADVERSE EVENTS:
Time Frame: 12 week treatment period plus 30 days after the last dose.
Description: Adverse events (AEs)were collected from the time of signing informed consent to the study and followup period (30 days). AEs were observed by the investigator (Inv) or reported by the participant. The nature of the event, time of onset, duration and intensity were documented together with the Inv assessment of the causal relationship to the drug.
Groups:
- Amlodipine 5 mg; Amlodipine 5mg and Olmesartan 20 mg; Amlodipine 5mg and Olmesartan 40 mg; Amlodipine 10 mg and Olmesartan 40 mg: All eligible participants began the active treatment period with amlodipine (Aml) 5 mg for Weeks 1-3. If blood pressure was greater than 120/80 at the end of 3 weeks, participants were titrated to the next regimen for weeks 4-6, and so on for weeks 7-9 and 10-12.
Arm/Group | Amlodipine 5 mg | Amlodipine 5mg and Olmesartan 20 mg | Amlodipine 5mg and Olmesartan 40 mg | Amlodipine 10 mg and Olmesartan 40 mg
Serious Adverse Events (participants affected / at risk) | 0/185 | 0/180 | 1/161 | 1/134
Other Adverse Events (participants affected / at risk) | 8/185 | 23/180 | 11/161 | 12/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amlodipine 5 mg (N=185) | Amlodipine 5mg and Olmesartan 20 mg (N=180) | Amlodipine 5mg and Olmesartan 40 mg (N=161) | Amlodipine 10 mg and Olmesartan 40 mg (N=134)
Limb amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 | 0 (0)
Transient ischemic attack (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Amlodipine 5 mg (N=185) | Amlodipine 5mg and Olmesartan 20 mg (N=180) | Amlodipine 5mg and Olmesartan 40 mg (N=161) | Amlodipine 10 mg and Olmesartan 40 mg (N=134)
Dizziness (Nervous system disorders) | 2 | 3 | 2 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 3
Nasopharyngitis (Infections and infestations) | 1 | 9 | 2 | 5
Oedema Peripheral (General disorders) | 3 | 5 | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 4 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"If identified by Daiichi Sankyo, Inc. (DSI), any of DSI's confidential information as defined herein shall be deleted…Nothing in this publication section shall be taken as giving DSI any right of editorial control over any publication prepared by Study Site."